CLINICAL TRIAL: NCT00552760
Title: A Double-Blind, Randomized, Placebo-Controlled Trial of Ramelteon for the Treatment of Insomnia and Mood Stability in Patients With Euthymic Bipolar Disorder.
Brief Title: Ramelteon for the Treatment of Insomnia and Mood Stability in Patients With Euthymic Bipolar Disorder
Acronym: Ram-TIME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Edward R. Norris, MD, Physician-Investigator, Lehigh Valley Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-006R
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramelteon (Experimental): 8 mg
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — one 8 mg tablet at bedtime for up to 6 months
  Other Names: Rozerem
  Arms: Ramelteon
Drug: Placebo — one tablet at bedtime for up to 6 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether treating sleep difficulties in patients with bipolar disorder also improves their mood stability.

DETAILED DESCRIPTION:
Patients with euthymic bipolar disorder, although free of significant mood symptoms, often have continued sleep disturbances. Improving patients' sleep by also normalizing the circadian rhythm will lead to fewer mood exacerbations. Ramelteon offers a new and more pharmacologically exact mechanism to re-synchronize the SCN. The administration of ramelteon for bipolar patients will improve sleep and will cause fewer mood exacerbations.

Patients with bipolar disorder often experience frequent mood alterations that are attempted to be controlled by mood stabilizing agents and anti-psychotic agents. Both classes of medications have numerous significant side effects. Establishing that ramelteon is helpful in the sleep of patients with bipolar disorder and helpful in mood stability will increase the number of treatment options for bipolar patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent before initiation of any study-related procedures
2. Men and women aged 18 to 65 years.
3. A documented clinical diagnosis according to the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision) meeting criteria 296.4x Bipolar I disorder, most recent episode manic, 296.6x Bipolar I disorder, most recent episode mixed, or 296.5x Bipolar I disorder, most recent episode depressed.
4. PSQI total score of >=5.
5. MADRS total score of <=12.
6. YMRS total score of <= 12
7. Female patients of childbearing potential must have a negative urine pregnancy test at enrollment and be willing to use a reliable method of birth control, i.e., double-barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device or tubal ligation, during the study.
8. Be able to understand and comply with the requirements of the study, as judged by the investigator.
9. Outpatient status at enrollment.

Exclusion Criteria:

1. Patients with a diagnosis of DSM-IV Axis II disorder which has a major impact on the patient's current psychiatric status.
2. Presence of prohibited medications of antidepressants (including MAOI's) and systemic corticosteroids.
3. Patients with a diagnosis of primary insomnia disorders
4. Patients with a diagnosis of severe chronic obstructive pulmonary disease
5. A clinical finding that is untreated (eg, hypertension, poorly controlled diabetes, angina) or that, in the opinion of the investigator, would be negatively affected by the study medication or that would affect the study medication.
6. Patients with active substance abuse diagnoses (except tobacco abuse).
7. Known history of intolerance or hypersensitivity to ramelteon or to any other component in the tablet.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward R. Norris, MD, Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Hospital, Department of Psychiatry, Allentown, Pennsylvania, United States

REFERENCES:
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Dokucu ME, Yu L, Taghert PH. Lithium- and valproate-induced alterations in circadian locomotor behavior in Drosophila. Neuropsychopharmacology. 2005 Dec;30(12):2216-24. doi: 10.1038/sj.npp.1300764. PMID 15956996
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Jones SH, Hare DJ, Evershed K. Actigraphic assessment of circadian activity and sleep patterns in bipolar disorder. Bipolar Disord. 2005 Apr;7(2):176-86. doi: 10.1111/j.1399-5618.2005.00187.x. PMID 15762859
- [Background] American Psychiatric Association: Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision. Washington, CD, American Psychiatric Association, 2000.
- [Result] Norris ER, Karen Burke, Correll JR, Zemanek KJ, Lerman J, Primelo RA, Kaufmann MW. A double-blind, randomized, placebo-controlled trial of adjunctive ramelteon for the treatment of insomnia and mood stability in patients with euthymic bipolar disorder. J Affect Disord. 2013 Jan 10;144(1-2):141-7. doi: 10.1016/j.jad.2012.06.023. Epub 2012 Sep 7. PMID 22963894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in October 2007 and was completed by August 2009. Participants, who at the time were receiving outpatient psychiatric services through Lehigh Valley Hospital, were recruited via referral through the department of psychiatry, and also through print advertisement. Participants received a $20 travel stipend for each appointment.
Pre-assignment Details: 90 participants signed the informed consent document, 7 were screen failures, and 83 were randomized to receive either Ramelteon or placebo. During the study, both groups were maintained on their usual medications for bipolar disorder and were not allowed to have any meds changed, as this would signify a manic or depressed event.
Period: Overall Study
Arm/Group | Ramelteon | Placebo
Started | 42 | 41
Completed | 16 | 8
Not Completed | 26 | 33
Not completed — Adverse Event | 3 | 5
Not completed — Relapsed- Depressed Event | 10 | 16
Not completed — Relapse- Manic Event | 3 | 3
Not completed — Relapsed- Mixed Event | 3 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Non-compliance | 1 | 1
Not completed — Medical Condition | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Medication Change | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon | Placebo | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 41 | 83
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.0) | 45.2 (10.8) | 45.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 16 | 15 | 31
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI) Global Score
Description: Self-rated scale to measure quality of sleep via questions regarding sleep latency, duration, efficiency, disturbances, use of sleep medication, and daytime dysfunction. Scores range from 0-21, higher scores represent more significant sleep disturbance.
Time Frame: Monthly for 6 months
Population: Intent to Treat Analysis; excludes 7 screen failures.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 42 | 41
units on scale
  Baseline | 10.17 (0.53) | 10.88 (0.53)
  Month 1 | 8.16 (0.56) | 9.28 (0.57)
  Month 2 | 7.93 (0.63) | 9.71 (0.64)
  Month 3 | 7.89 (0.68) | 10.38 (0.78)
  Month 4 | 7.21 (0.62) | 9.03 (0.75)
  Month 5 | 6.62 (0.59) | 8.66 (0.77)
  Month 6 | 6.90 (0.72) | 8.76 (0.98)

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: 10-item, standardized, well-validated scale used to measure severity of depressive symptoms; sensitive to treatment effects in depressed outpatients. Scores range from 0-60, higher scores represent more severe depressive symptoms.
Time Frame: Monthly for 6 months
Population: Intent to Treat Analysis; excludes 7 screen failures
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 42 | 41
units on scale
  Baseline | 7.79 (0.42) | 8.27 (0.43)
  Month 1 | 8.34 (0.67) | 8.90 (0.68)
  Month 2 | 7.23 (0.84) | 11.13 (0.85)
  Month 3 | 9.17 (1.00) | 11.85 (1.24)
  Month 4 | 8.45 (1.05) | 13.03 (1.39)
  Month 5 | 8.56 (1.24) | 11.59 (1.73)
  Month 6 | 10.40 (1.48) | 10.46 (2.18)

3. Secondary Outcome: Young Mania Rating Scale (YMRS) Total Score
Description: 11-item standardized, well-validated scale used to measure manic symptoms; sensitive to treatment effects in manic patients. Scores range from 0-60, higher scores represent more severe manic symptoms.
Time Frame: Monthly for 6 months
Population: Intent to Treat Analysis; excludes 7 screen failures
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 42 | 41
units on scale
  Baseline | 7.02 (0.43) | 6.59 (0.44)
  Month 1 | 5.89 (0.51) | 6.46 (0.52)
  Month 2 | 5.91 (0.80) | 7.75 (0.82)
  Month 3 | 6.60 (0.84) | 8.09 (1.00)
  Month 4 | 5.93 (0.70) | 4.95 (0.93)
  Month 5 | 5.18 (0.65) | 5.71 (0.88)
  Month 6 | 6.51 (1.00) | 6.72 (1.35)

4. Secondary Outcome: Clinical Global Impressions Bipolar Version(CGI-BP) Severity of Illness Overall Score
Description: 3-part (mania, depression, overall bipolar illness), physician-administered scale used to assess global illness severity; used to measure change. Each part is rated from 1-7, higher scores represent more severe mental illness. Only overall bipolar rating was used.
Time Frame: Monthly for 6 months
Population: Intent to Treat Analysis; excludes 7 screen failures
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 42 | 41
units on scale
  Baseline | 2.14 (0.13) | 2.15 (0.13)
  Month 1 | 2.29 (0.15) | 2.25 (0.15)
  Month 2 | 2.24 (0.18) | 2.90 (0.19)
  Month 3 | 2.53 (0.22) | 2.93 (0.27)
  Month 4 | 2.36 (0.21) | 2.98 (0.29)
  Month 5 | 2.46 (0.23) | 2.99 (0.34)
  Month 6 | 2.54 (0.23) | 2.41 (0.34)

5. Secondary Outcome: Cumulative Proportion of Participants in Each Arm Surviving Without Relapse
Description: Survival analysis techniques, including Kaplan Meier curves, were used to evaluate group differences in time to relapse. Relapse was defined as a medication initiation or change for manic/depressed/mixed symptoms, a hospitalization for manic/depressed/mixed symptoms, MADRS score >= 16, YMRS score > 14, and suicide risk or imminent risk of suicide. Time to relapse was measured discretely in terms of the number of assessment visits until discontinued from the study.
Time Frame: Monthly for 6 months
Population: Intent to Treat Analysis; excludes 7 screen failures.
Measure: Number; unit: Cumulative proportion of participants
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 42 | 41
Cumulative proportion of participants
  Baseline | 1.00 | 1.00
  Month 1 | 0.929 | 0.951
  Month 2 | 0.849 | 0.588
  Month 3 | 0.716 | 0.448
  Month 4 | 0.661 | 0.384
  Month 5 | 0.632 | 0.320
  Month 6 | 0.566 | 0.320

ADVERSE EVENTS:
Arm/Group | Ramelteon | Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 12/42 | 12/41
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramelteon (N=42) | Placebo (N=41)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Diarrhea NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (4)
Forgetfulness (General disorders) | 0 (0) | 1 (1)
Headache NOS (General disorders) | 1 (1) | 1 (1)
Insomnia exacerbated (General disorders) | 1 (1) | 0 (0)
Restless legs (General disorders) | 0 (0) | 1 (1)
Somnolence (General disorders) | 3 (3) | 1 (1)
Vivid dreams (General disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes